CLINICAL TRIAL: NCT04315493
Title: A Randomized, Open, Single-dose, Two-cycle, Double-sequence, Crossover Study to Investigate the Effects of a Low-fat Diet On the Pharmacokinetics of Healthy Chinese Adult Participants After Oral Administration of Pyrotinib Maleate Tablets
Brief Title: Effect of Low-fat Diet on the Pharmacokinetics of Pyrotinib in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BLTN-If
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Diet, Fat-Restricted; P-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: pyrotinib maleate fasted in P1, low-fat diet in P2
- B (Experimental)
  Interventions: Drug: pyrotinib maleate low-fat diet in P1, fasted in P2

INTERVENTIONS:
Drug: pyrotinib maleate fasted in P1, low-fat diet in P2 — pyrotinib maleate administration in fasted condition in period 1, pyrotinib maleate administration after low-fat diet in period 2
  Arms: A
Drug: pyrotinib maleate low-fat diet in P1, fasted in P2 — pyrotinib maleate administration after low-fat diet in period 1, pyrotinib maleate administration in fasted condition in period 2
  Arms: B

SUMMARY:
The primary objective of the study is to evaluate the effect of low-fat diet on pharmacokinetics of healthy Chinese adult participants after oral administration of pyrotinib maleate tablets.

The secondary objective of the study is to evaluate the safety of single dose of pyrotinib orally in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
4. Have no fertility plan and agree to adopt effective contraceptive measures within 2 weeks before the first study drug administration and up to 3 months after the last study drug administration. Negative pregnancy test for women of child-bearing age before the first study drug administration;
5. Male body weight ≥ 50kg, female body weight ≥ 45kg, and body mass index (BMI) within the range of 19 ~ 26 kg/m^2 (including 19 and 26);
6. During screening period, the comprehensive physical examination (vital signs and physical examination), routine laboratory examination (blood routine, urine routine, blood biochemistry, coagulation,etc), 12-lead electrocardiogram (ECG), chest X-ray, cardiac ultrasound, B ultrasound and other examination results must be within the normal range, or judged to be "no clinical significance (NCS)" if beyond the normal range;

Exclusion Criteria:

1. Blood donation within 3 months before the first drug administration and blood loss greater than 400 mL, or receiving blood transfusion;
2. Allergic constitution, including those with severe drug allergies or a history of drug allergies, or known allergy to the research drug;
3. History of drug use, or drug abuse screening positive; history of drug abuse within the past five years or have used drugs 3 months before the test;
4. Alcoholic or often drinkers (the average drinking amount is more than 14 units a week: 1 unit= 285 ml beer or 45 ml spirits or 100 ml wine; ≥5 cigarettes per day) and can't quit smoking and alcohol during the study; alcohol test positive;
5. The 12-lead ECG with female QTcF > 470ms or male QTcF > 450ms;
6. Left ventricular ejection fraction (LVEF) <50% by echocardiography;
7. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.
8. Those who have undergone any surgery within 6 months before screening;
9. Those who have taken hepatotoxic drugs (such as dapsone, erythromycin, fluconazole, ketoconazole, rifampicin) for a long time within the 6 months before screening;
10. Those who have taken any research drugs within 3 months before the first drug administration;
11. Use any drugs that changes liver enzyme activity within 4 weeks before the first drug administration;
12. Use any prescription or over-the-counter drug, any vitamin product, health supplement or herbal medicine within 2 weeks prior to first drug administration;
13. Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases;
14. HCV antibody positive, HIV antibody positive, HBsAg positive, and syphilis antibody positive;
15. Consumption of grapefruit or grapefruit-containing products, foods or beverages containing caffeine, xanthine, or alcohol within 48 hours before the first drug administration; strenuous exercise or other factors that effect on drug absorption, distribution, metabolism and excretion;
16. Have special requirements on diet and cannot comply with the diet and corresponding regulations provided by the test;
17. History of dizzy needles or blood dizziness; difficulty in venous blood collection or inability to tolerate venipuncture;
18. lactating women;
19. Other factors that are not suitable for participating in the study, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of pyrotinib | through study completion, an average of 28 days
  Peak Plasma Concentration (Cmax) of pyrotinib
Pharmacokinetics parameter: AUC of pyrotinib | through study completion, an average of 28 days
  Area under the plasma concentration versus time curve (AUC) of pyrotinib

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of pyrotinib | through study completion, an average of 28 days
  Time of maximum observed concentration (Tmax) of pyrotinib
Pharmacokinetics parameter: T1/2 of pyrotinib | through study completion, an average of 28 days
  Half time (T1/2) of pyrotinib
Pharmacokinetics parameter: CL/F of pyrotinib | through study completion, an average of 28 days
  Total body clearance for extravascular administration (CL/F) of pyrotinib
Pharmacokinetics parameter: Vz/F of pyrotinib | through study completion, an average of 28 days
  Volume of distribution (Vz/F) of pyrotinib
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 28 days
  An adverse event is any untoward medical occurrence in a patient or clinical study participant

IPD SHARING:
Plan to Share IPD: No